CLINICAL TRIAL: NCT03674892
Title: Assessing the Efficacy of Intranasal Neurostimulation in Ameliorating Symptoms of Neuropathic Corneal Pain
Brief Title: Intranasal Neurostimulation in Ameliorating Symptoms of Neuropathic Corneal Pain
Acronym: INSTANT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original device is now discontinued; we are changing the study device shortly
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12978
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cornea
Keywords: Intranasal Neurostimulation
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: non-randomized, open-label, single arm pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TrueTear™ intranasal neurostimulator (ITN) (Experimental): TrueTear™ intranasal neurostimulator (ITN)
  Interventions: Device: TrueTear™ intranasal neurostimulator (ITN)

INTERVENTIONS:
Device: TrueTear™ intranasal neurostimulator (ITN) — TrueTear™ intranasal neurostimulator (ITN)

SUMMARY:
This study is a prospective, interventional, open-label, single arm, non-randomized trial treating 30 patients with peripheral or mixed neuropathic corneal pain at their baseline exam and following 45 days and 90 days of daily use with the TrueTear™ ITN device.

DETAILED DESCRIPTION:
The investigators hypothesize that the stimulation through the ethmoidal nerve in the nasal cavity may have an inhibitory effect on the primary TG interneurons and block the ocular pain signaling to the brain.

The investigators propose a non-randomized, open-label, single arm pilot trial for treatment of neuropathic corneal pain (NCP) with ITN with the following specific aims:

Specific Aims:

1. To elucidate the efficacy of ITN in ameliorating pain among neuropathic corneal pain patients.
2. To elucidate the safety, efficacy, longevity of ITN in ameliorating pain among neuropathic corneal pain patients during a 90-day period with daily use.
3. To assess quality of life changes by treating neuropathic corneal pain with ITN during a 90-day period with daily use.

ELIGIBILITY:
Inclusion Criteria:

1. Age >22
2. Ability to consent to study.
3. Symptoms of neuropathic corneal pain for at least 3 months, such as burning, stinging, light sensitivity, discomfort or pain.
4. Positive in vivo confocal microscopy (IVCM) findings for NCP such as presence of microneuromas and decreased nerve density.
5. Fifty percent or more relief of pain or discomfort after instillation of Proparacaine eye drops as measured by the Visual Analogue Scale (VAS).

Exclusion Criteria:

1. Clinically significant acute ocular surface diseases, such as active infectious keratitis or recent ocular surgery in the past 3 months.
2. Chronic or recurrent epistaxis, coagulation disorders.
3. Nasal or sinus surgery or significant trauma to the nose.
4. Severe nasal airway obstruction or vascularized nasal polyps.
5. Cardiac demand pacemaker, implanted defibrillator, or other implanted electronic device in the head or neck.
6. Chronic or recurrent nosebleeds
7. Bleeding disorder
8. Known hypersensitivity (allergy) to the hydrogel material
9. Disabling arthritis, neuropathy, or limited motor coordination affecting self-handling of the device.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As outlined in the study protocol, this trial aimed to enroll 45 patients with neuropathic corneal pain and evaluate them at 45 and 90 days following daily use of the TrueTear™ device. However, due to the COVID-19 pandemic and related concerns about infection, only 21 patients enrolled in the study and completed the first visit. As this was a single arm study, all participants were assigned to the TrueTear™ intranasal neurostimulator (ITN) group.
Groups:
- Experimental: TrueTear™ Intranasal Neurostimulator (ITN): The TrueTear® ITN, recently approved by the FDA, is a portable neuromodulation device that delivers a small electrical current to the sensory nerves in the nasal cavity that stimulates the nasolacrimal reflex (NLR).
Period: Overall Study
Arm/Group | Experimental: TrueTear™ Intranasal Neurostimulator (ITN)
Started | 21
Month 1 Visit 3 | 12
Completed | 6
Not Completed | 15
Not completed — Lack of Efficacy | 5
Not completed — Lost to Follow-up | 3
Not completed — Migraine | 2
Not completed — Excessive Tearing | 1
Not completed — Increased Eye Pain | 1
Not completed — Increased Facial Pain | 1
Not completed — Sinus Irritation | 1
Not completed — Sinus Infection | 1

BASELINE CHARACTERISTICS:
Arm/Group | TrueTear™ Intranasal Neurostimulator (ITN)
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.05 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21
Randomly Selected Eye for Analysis (Right eye/Left eye) [Count of Participants; unit: Participants]
  Right eye OD | 11
  Left eye OS | 10
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: logMAR] | 0.09 (0.10)
Schirmer [Mean (Standard Deviation); unit: millimeters] — The Schirmer test was performed by placing a narrow filter-paper strip (5 x 35 mm strip of Whatman #41 filter paper) in the inferior cul-de-sac. The subject should gently close their eyes until five minutes have elapsed and the strips are removed. Aqueous tear production was measured by the length in millimeters that the strip wets during 5 minutes. The Schirmer test results range from 0 to 35 mm, with lower values indicating more severe dry eye.
  millimeters | 8.71 (7.00)
Tear Break Up Time [Mean (Standard Deviation); unit: seconds] | 6.70 (2.69)
Corneal Staining Score [Mean (Standard Deviation); unit: scores on a scale] — Corneal Staining Score: The NEI (National Eye Institute) corneal staining score is a standardized method used to assess the extent of corneal epithelial damage, typically visualized with fluorescein dye under cobalt blue light. The cornea is divided into five equal zones. Each zone is graded on a scale from 0 to 3, based on the number and density of punctate epithelial erosions (staining spots). The scores from all five zones are summed (0-15), giving a total corneal staining score. Higher scores indicates more severe dryness.
  scores on a scale | 2.56 (4.03)
Conjunctival Staining Score [Mean (Standard Deviation); unit: Scores on a scale] — The NEI (National Eye Institute) conjunctival staining score is used to assess damage or dryness-related staining of the bulbar conjunctiva by using lissamine green. The exposed bulbar conjunctiva is divided into six regions. Each zone is scored from 0 to 3, The scores for all six zones are summed, giving a total conjunctival staining score. The conjunctival staining score ranges from 0 to 18, with higher scores indicating more severe dry eye.
  Scores on a scale | 2.44 (4.03)
Intraocular Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 13.76 (3.22)
Proparacaine Challenge Test [Mean (Standard Deviation); unit: Units on a scale] — Patients marked their current pain intensity on a 10 cm horizontal visual analogue scale (VAS), with 'no pain' (0) at the left end and 'worst imaginable pain' (10) at the right end. This score was recorded as centimeter and given as 'before'. One drop of Proparacaine was then topically applied, and after 90 seconds, patients marked their pain intensity on the same scale. This second score was recorded and given as 'after'. The pain scale ranges from 0 to 10, with higher scores indicating greater pain severity.
  Units on a scale
    Before | 5.80 (3.08)
    After | 1.80 (1.54)
Proparacaine Challenge Test Percent Change [Mean (Standard Deviation); unit: percentage change] — The mean post-instillation pain intensity was subtracted from the mean pre-instillation value, divided by the mean pre-instillation intensity, and multiplied by 100 to calculate the percentage of pain change following proparacaine eyedrop instillation. Values range from -100 to 0; a value of -100 indicates that corneal pain originated entirely from peripheral corneal nerves, whereas 0 indicates that the pain originated entirely from non-ocular surface sources, such as the trigeminal ganglion or the upstream central nervous system.
  percentage change | -68.96 (19.12)
Cold Saline Test [Mean (Standard Deviation); unit: units on a scale] — Patients marked their current pain intensity on a 10 cm horizontal visual analogue scale (VAS), with 'no pain' (0) at the left end and 'worst imaginable pain' (10) at the right end. This score was recorded in centimeter and given as 'before'. One drop of cold 0.9% preservative-free saline was then topically applied, and immediately after patients marked their pain intensity on the same scale. This second score was recorded and given as 'after'. Higher scores indicate greater pain severity.
  units on a scale
    Before | 4.40 (2.21)
    After | 2.75 (2.24)
Hypertonic Test [Mean (Standard Deviation); unit: units on a scale] — Patients marked their current pain intensity on a 10 cm horizontal visual analogue scale (VAS), with 'no pain' (0) at the left end and 'worst imaginable pain' (10) at the right end. This score was recorded in centimeters and designated as 'before'. One drop of 5% sodium chloride (Muro 128®) was then topically applied, and after twenty seconds, patients marked their pain intensity on the same scale. This second score was recorded and designated as 'after'. The pain scale ranges from 0 to 10, with higher scores indicating greater pain severity.
  units on a scale
    Before | 3.30 (2.79)
    After | 5.25 (3.53)
Neuropathic Corneal Pain Type [Count of Participants; unit: Participants] — One drop of Proparacaine Hydrochloride Ophthalmic Solution 0.5% was topically applied in both eyes to differentiate between the peripheral versus central component of the patient's eye pain or discomfort. The level of discomfort/pain was then assessed by the visual analogue scale (VAS) questionnaire. Patients who experienced complete eye pain relief after proparacaine instillation were classified as having peripheral neuropathic corneal pain, whereas those with partial relief were classified as having mixed neuropathic corneal pain.
  Participants
    Peripheral | 16
    Mixed | 5
Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Patients marked their current pain intensity on a 10 cm horizontal visual analogue scale, with 'no pain' (0) at the left end and 'worst imaginable pain' (10) at the right end. This score was recorded as 'Pre-stimulation'. Each participant was asked to apply the intranasal neurostimulation device for 1 minute, and if no change in discomfort is noted, to continue for up to 3 minutes. Then patients marked their pain intensity on the same scale and recorded as 'Post-stimulation'. The pain scale ranges from 0 to 10, with higher scores indicating greater pain severity.
  units on a scale
    Pre-stimulation | 5.73 (2.09)
    Post-stimulation | 1.92 (1.67)
    Difference | -3.81 (1.88)
Pain Intensity Change Percent after Intranasal Neurostimulation [Mean (Standard Deviation); unit: percent change] — Pain Intensity Change Percent after Intranasal Neurostimulation was calculated by subtracting the mean post-stimulation pain intensity from the mean pre-stimulation value, then dividing by the mean pre-stimulation intensity and multiplying by 100 to obtain the percentage change. Values ranged from -100 to 100, with higher values indicating less pain reduction or pain increase after intranasal neurostimulation and a worse outcome.
  percent change | -66.49 (29.38)
Ocular Surface Disease Index (OSDI) Score [Mean (Standard Deviation); unit: Scores on a scale] — The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire, with each question scored on a scale from 0 to 4, where 0 indicates 'none of the time' and 4 indicates 'all of the time.' To calculate the OSDI score, the sum of the scores from all answered questions was multiplied by 25 and then divided by the total number of questions answered. OSDI scores range from 0 to 100, with higher scores indicating more severe ocular surface symptoms and a worse outcome.
  Scores on a scale | 69.96 (19.83)
Ocular Surface Disease Index (OSDI) Dimensions [Mean (Standard Deviation); unit: Scores on a scale] — (0 = None of the time, 1 = Some of the time, 2 = Half of the time, 3 = Most of the time, 4 = All of the time)
  Scores on a scale
    Light Sensitivity | 2.85 (1.56)
    Gritty | 2.37 (1.30)
    Painful Eyes | 3.30 (0.86)
    Blurred Eyes | 2.30 (1.49)
    Poor Vision | 2.26 (1.36)
    Reading | 2.61 (0.97)
    Driving Night | 2.50 (1.54)
    Working ATM/Computer | 3.11 (1.13)
    Watching TV | 2.94 (2.01)
    Windy Conditions | 3.17 (1.15)
    Low Humidity | 3.53 (0.62)
    Areas with Air Conditioner | 3.64 (0.63)
Ocular Pain Assessment Survey (OPAS) Dimensions [Mean (Standard Deviation); unit: Scores on a scale] — The overall severity of pain (0 = no pain, 10 = worst pain ever)
  Scores on a scale
    Overall Pain | 5.50 (2.42)
    Most Eye Pain Intensity in the past 24 hours | 7.87 (1.99)
    Least Eye Pain Intensity in the past 24 hours | 3.21 (2.10)
    Average Eye Pain Intensity in the past 24 hours | 5.75 (1.96)
    Most Eye Pain Intensity in the past 2 weeks | 7.82 (2.02)
    Least Eye Pain Intensity in the past 2 weeks | 4.00 (2.29)
    Average Eye Pain Intensity in the past 2 weeks | 5.65 (1.96)
    Non-Eye Pain in the past 24 hours | 4.68 (3.64)
    Non-Eye Pain in the past 2 weeks | 5.42 (3.92)
Ocular Pain Assessment Survey (OPAS) [Mean (Standard Deviation); unit: The percentage of time (%)] — The percentage of time spent thinking about non-eye pain (face/head) (0% = Not at all, 100% = All the time)
  The percentage of time (%) | 46.68 (36.90)
Ocular Pain Assessment Survey (OPAS) Quality of Life Parameters [Mean (Standard Deviation); unit: Scores on a scale] — How much pain has interfered with/affected the following (0 = Not at all, 10 = Completely)
  Scores on a scale
    Reading | 7.37 (2.88)
    Driving | 6.50 (3.31)
    General activity (walking, doing house chores) | 5.52 (3.31)
    Mood | 7.00 (2.45)
    Sleep | 4.55 (3.28)
    Enjoying Life/ Relations with other people | 6.65 (3.26)
Ocular Pain Assessment Survey (OPAS) Quality of Life Parameters [Mean (Standard Deviation); unit: The percentage of time (%)] — The final dimension of the Ocular Pain Assessment Survey's Quality of Life section assesses the percentage of time the patient spends thinking about eye pain. Scores range from 0 to 100, with higher scores indicating more time spent thinking about eye pain and greater pain severity.
  The percentage of time (%) | 74.12 (27.90)
Ocular Pain Assessment Survey (OPAS) Average Quality of Life (QoL) Score: [Mean (Standard Deviation); unit: Scores on a scale] — The Quality of Life (QoL) section of Ocular Pain Assessment Survey (OPAS) includes 7 items: the first 6 are rated on a 0-10 scale, while the last item is scored as a percentage (0-100). To calculate the average OPAS QoL score, the percentage-based item is first converted to a 0-10 scale. Then, the sum of all answered item scores is divided by the total number of items completed. OPAS Average QoL scores range from 0 to 10, with higher scores indicating greater interference of daily activities due to ocular surface symptoms, lower QoL, and a worse outcome.
  Scores on a scale | 6.46 (2.48)
Ocular Pain Assessment Survey (OPAS) Aggravating Factors [Mean (Standard Deviation); unit: percent (%)] — How much pain is increased when exposed to the following factors (0% = No change, 100% = Severe increase)
  percent (%)
    Wind, dry air, heat, air conditioning | 79.72 (32.47)
    Volatile chemicals (cleaning agents, fumes, cosmetic) | 65.00 (38.17)
Ocular Pain Assessment Survey (OPAS) Associated Factors [Mean (Standard Deviation); unit: percent (%)] — How often eye pain is accompanied by the following symptoms (0% = Never, 100% = All the time)
  percent (%)
    Redness | 50.26 (34.74)
    Burning | 73.00 (25.15)
    Sensitivity to light | 75.25 (36.65)
    Tearing | 38.95 (36.99)
Ocular Pain Assessment Survey (OPAS) Symptom Relief [Mean (Standard Deviation); unit: percent (%)] — Pain relief experienced since last visit (0% = No relief, 100% = Complete relief)
  percent (%)
    Eye Pain | 33.63 (23.03)
    Non-Eye Pain (face/head) | 23.75 (27.61)
Impact of Dry Eye in Everyday Life (IDEEL) Daily Activities [Mean (Standard Deviation); unit: Scores on a Scale] — The IDEEL questionnaire is a 57-item instrument and comprises three modules: dry eye impact on daily life, dry eye treatment satisfaction, and dry eye symptom bothers. In this study, the dry eye impact on daily life module was used, which consists of 27 items and assesses Quality of Life (QoL) in three aspects over the previous two weeks: daily activities, feelings, and work. Aside from the yes-or-no questions, the other questions are answered on a 0-5 Likert scale, where zero signifies an inability to perform the activity. Lower scores indicate more severe disability and worse outcome.
  Scores on a Scale
    Doing close work in the morning or afternoon | 2.60 (1.59)
    Doing close work in the evening or at night | 2.73 (1.43)
    Driving | 3.35 (1.64)
    Being around and/or using scented products | 3.21 (1.96)
    Working on a computer | 2.46 (1.68)
    Going somewhere where there is tobacco smoke | 2.40 (1.91)
    Wearing contact lenses | 3.92 (2.05)
    Wearing make-up | 2.57 (1.86)
    Flying on an airplane | 3.53 (1.71)
Impact of Dry Eye in Everyday Life (IDEEL) Feelings [Mean (Standard Deviation); unit: Scores on a Scale] — How often feelings are had because of dry eyes over the last two weeks (1 = All of the time, 2 = Most of the time, 3 = Some of the time, 4 = A little of the time, 5 = None of the time)
  Scores on a Scale
    Irritability | 1.73 (1.03)
    Impatience | 2.13 (1.12)
    Feeling sad | 1.80 (1.20)
    Worry that my dry eyes will get worse | 1.33 (1.32)
    Feeling annoyed | 1.93 (1.22)
    Feeling like my eyes do not look nice | 1.66 (1.44)
    Feeling like I have to make adjustments to my life | 1.06 (1.12)
    Feeling different from other people | 1.66 (1.63)
    Feeling like I am always aware of my eyes | 0.80 (1.08)
    Feeling older than I really am | 2.00 (1.64)
    Feeling like people look at me and think I am fine when I'm not | 1.73 (1.66)
    Feeling like there is nothing I can do for my dry eyes | 1.26 (1.38)
Impact of Dry Eye in Everyday Life (IDEEL) Work [Count of Participants; unit: Participants]
  Yes | 10
  No | 5
  No answer | 6
Impact of Dry Eye in Everyday Life (IDEEL) Situations at Work [Mean (Standard Deviation); unit: IDEEL Score] — How often were the following situations experienced over the last two weeks at work because of dry eyes? (0 = All of the time, 1 = Most of the time, 2 = Some of the time, 3 = A little of the time, 4 = None of the time)
  IDEEL Score
    Feeling distracted | 1.64 (1.00)
    Feeling like I couldn't concentrate | 1.71 (1.06)
    Having to take a break from work | 1.38 (1.12)
    Having to change the way I work | 1.28 (1.26)
    Having to change my work environment | 1.28 (1.58)
Filter Glasses Test [Mean (Standard Deviation); unit: Units on a scale (0-100)] — This test was done in a dimly lit room and each eye was assessed separately. The other eye was covered with an occluder to eliminate exposure to the light. The study eye was covered using a 100% opaque filter, and then the opacity of the filters was reduced in decrements of 10%. Ten graded filters were developed for this purpose; starting with the 100% opaque filter, the filter at which the patient started to feel pain/photophobia was noted. Values range 0-100; higher opacity filters reflect more photosensitivity and a worse outcome.
  Units on a scale (0-100) | 78.00 (8.36)

OUTCOME MEASURES:

1. Primary Outcome: Change to Overall Pain by the Visual Analogue Scale (VAS) After Intranasal Neurostimulator (ITN) Stimulation at Baseline
Description: The Visual Analogue Scale (VAS) is a 10 cm line, with one end labeled 'no pain' (which is equivalent to a score of 0 on the numerical scale) and the other end labeled 'worst pain imaginable' (which is equivalent to a score of 10 on the numerical scale). The patient is asked to mark the scale according to the intensity of their eye pain, and the examiner measures the distance in centimeters from the 'no pain' end of the line to score the VAS. The level of discomfort/pain before and after ITN was assessed using the VAS questionnaire (0-10). The changes in overall eye pain after ITN were recorded. Higher scores on the VAS indicate more intense pain and a worse outcome.
Time Frame: immediately before and after ITN on Day 1 (baseline)
Population: Post-stimulation minus pre-stimulation pain scores of all patients who underwent intranasal neurostimulation at the 1-day (baseline) visit.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients Participated Baseline Visit: Difference of pain scores before and after ITNS at baseline visit
  ITNS:Intranasal neurostimulation with TrueTear™ intranasal neurostimulator (ITN)
Arm/Group | All Patients Participated Baseline Visit
Number analyzed (Participants) | 21
score on a scale | -3.81 (0.41)

2. Secondary Outcome: Change to Overall Pain by the Visual Analogue Scale (VAS) After Daily Intranasal Neurostimulator (ITN) Stimulation Over 45-day Period
Description: The VAS is a 10 cm line, with one end labeled 'no pain' (which is equivalent to a score of 0 on the numerical scale) and the other end labeled 'worst pain imaginable' (which is equivalent to a score of 10 on the numerical scale). The patient is asked to mark the scale according to the intensity of their eye pain, and the examiner measures the distance in centimeters or millimeters from the 'no pain' end of the line to score the VAS. The level of discomfort/pain before and after ITN was assessed using the VAS questionnaire (0-10). The changes in overall eye pain after ITN were recorded. Higher scores on the VAS indicate more intense pain and a worse outcome.
Time Frame: immediately before and after ITN on Day 45
Population: Post-stimulation minus pre-stimulation pain scores of all patients who underwent intranasal neurostimulation at the 45-day visit.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients Participated 45 Day Visit: Difference of pain scores before and after ITNS at 45 Day Visit
  ITNS:Intranasal neurostimulation with TrueTear™ intranasal neurostimulator (ITN)
Arm/Group | All Patients Participated 45 Day Visit
Number analyzed (Participants) | 12
score on a scale | -1.58 (0.39)

3. Secondary Outcome: Change to Overall Pain by the Visual Analogue Scale (VAS) After Daily Intranasal Neurostimulator (ITN) Stimulation Over 90-day Period
Description: The Visual Analogue Scale (VAS) is a 10 cm line, with one end labeled 'no pain' (which is equivalent to a score of 0 on the numerical scale) and the other end labeled 'worst pain imaginable' (which is equivalent to a score of 10 on the numerical scale). The patient is asked to mark the scale according to the intensity of their eye pain, and the examiner measures the distance in centimeters or millimeters from the 'no pain' end of the line to score the VAS. The level of discomfort/pain before and after ITN was assessed using the VAS questionnaire (0-10). The changes in overall eye pain after ITN were recorded. Higher scores on the VAS indicate more intense pain and a worse outcome.
Time Frame: immediately before and after ITN on Day 90
Population: Post-stimulation minus pre-stimulation pain scores of all patients who underwent intranasal neurostimulation at the 90-day visit.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients Participated 90 Day Visit: Difference of pain scores before and after ITNS at 90-day visit.
  ITNS:Intranasal neurostimulation with TrueTear™ intranasal neurostimulator (ITN)
Arm/Group | All Patients Participated 90 Day Visit
Number analyzed (Participants) | 6
score on a scale | -0.75 (0.83)

4. Secondary Outcome: Quality of Life as Measured With OPAS at Baseline
Description: The Ocular Pain Assessment Survey (OPAS) is a multidimensional questionnaire that assesses eye pain, non-eye pain, quality of life (QoL), aggravating factors, and associated factors. The QoL section evaluates seven dimensions, with the first six graded using numerical rating scales (0-10) and the final question expressed as a percentage (0-100). Higher scores indicate severe pain and lower QoL in the QoL section of OPAS questionnaire. Ranges: 0-10 for the "Reading and/or computer use", "Driving and/or watching TV", "General Activity", "Mood", "Sleep", "Enjoying Life/ Relationship. "Time spent thinking about pain" dimensions and 0-100. Higher scores indicate worse QoL.
Time Frame: Day 1 (Baseline)
Population: All Patients Participated 1 Day (Baseline) Visit
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients Participated Baseline Visit: Quality of life Scores as measured with Ocular Pain Assessment Survey at 1 day (baseline) Visit
Arm/Group | All Patients Participated Baseline Visit
Number analyzed (Participants) | 21
score on a scale
  Reading and/or computer use | 7.37 (0.64)
  Driving and/or watching tv | 6.50 (0.78)
  General activity | 5.52 (0.75)
  Mood | 7.00 (0.54)
  Sleep | 4.55 (0.77)
  Enjoying Life/Relationship | 6.65 (0.73)
  Time spent thinking about pain | 74.12 (6.76)

5. Secondary Outcome: Quality of Life as Measured Daily With OPAS at 45 Days
Description: as for outcome 4
Time Frame: 45 days
Population: All Patients Participated 45 Day Visit
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients Participated 45 Day Visit: Quality of life Scores as measured with Ocular Pain Assessment Survey at 45 Visit after daily intranasal neurostimulation treatment
Arm/Group | All Patients Participated 45 Day Visit
Number analyzed (Participants) | 12
score on a scale
  Reading and/or computer use | 5.50 (0.85)
  Driving and/or watching TV | 5.03 (0.96)
  General Activity | 4.03 (0.80)
  Mood | 5.42 (0.74)
  Sleep | 3.64 (0.90)
  Enjoying Life/ Relationship | 4.89 (0.70)
  Time spent thinking about pain | 59.6 (8.91)

6. Secondary Outcome: Quality of Life as Measured Daily With OPAS at 90 Days
Description: as for outcome 4
Time Frame: 90 days
Population: All Patients Participated 90 Day Visit
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients Participated 90 Day Visit: Quality of life Scores as measured with Ocular Pain Assessment Survey at 90 Visit after daily intranasal neurostimulation treatment
Arm/Group | All Patients Participated 90 Day Visit
Number analyzed (Participants) | 6
score on a scale
  Reading and/or computer use | 4.80 (1.82)
  Driving and/or watching TV | 5.00 (1.92)
  General activity | 2.50 (0.89)
  Mood | 4.40 (1.37)
  Sleep | 2.00 (1.37)
  Enjoying Life/ Relationship | 4.30 (1.57)
  Time spent thinking about pain | 53.31 (26.01)

7. Secondary Outcome: Overall Change in Quality of Life as Measured Daily With OPAS
Description: The Ocular Pain Assessment Survey (OPAS) is a multidimensional questionnaire that assesses eye pain, non-eye pain, quality of life (QoL), aggravating factors, and associated factors. The QoL section evaluates seven dimensions, with the first six graded using numerical rating scales (0-10) and the final question expressed as a percentage (0-100). Higher scores indicate severe pain and lower QoL in the QoL section of OPAS questionnaire.
  Percentage changes in the scores between baseline vs 45-day visit and baseline vs 90-day visit after daily intranasal neurostimulation are given below.
Time Frame: Baseline vs day 45 visit and Baseline vs day 90 visit
Population: Patients participated INSTANT study visits
Measure: Mean (Standard Error); unit: percent change
Groups:
- Baseline vs 45-day Visit: Percentage changes in the QoL scores between baseline and 45-day visit after daily ITN
  ITN: Intranasal neurostimulation with TrueTear™ intranasal neurostimulator QoL: Quality of life dimensions in ocular pain assessment questionnaire
- Baseline vs 90-day Visit: Percentage changes in the QoL scores between baseline and 90-day visit after daily ITN
  ITN: Intranasal neurostimulation with TrueTear™ intranasal neurostimulator QoL: Quality of life dimensions in ocular pain assessment questionnaire
Arm/Group | Baseline vs 45-day Visit | Baseline vs 90-day Visit
Number analyzed (Participants) | 12 | 6
percent change
  Reading and/or computer use | -25.37 (11.39) | -34.87 (17.72)
  Driving and/or watching TV | -22.61 (11.97) | -23.07 (19.32)
  General Activity | -26.99 (30.92) | -54.71 (15.02)
  Mood | -22.57 (9.20) | -37.14 (10.84)
  Sleep | -23.95 (30.32) | -56.04 (40.44)
  Enjoying life/ Relationship | -26.46 (13.94) | -35.33 (26.20)
  Time spent thinking about pain | -19.56 (34.50) | -28.07 (25.72)

8. Secondary Outcome: Percent Change From Pain Level Dimension Questions of the Ocular Pain Assessment Survey (OPAS)
Description: The Ocular Pain Assessment Survey (OPAS) is a multidimensional questionnaire that assesses eye pain, non-eye pain, quality of life (QoL), aggravating factors, and associated factors. Eye pain intensity was assessed using a numerical scale (0-10) for the most, least, and average pain in the past 24 hours and 2 weeks. Higher scores indicate severe pain of OPAS questionnaire. The percent changes in pain intensity between baseline vs 45-day and baseline vs 90-day are provided below.
Time Frame: Baseline vs day 45 visit and Baseline vs day 90 visit
Population: Patients participated INSTANT study visits
Measure: Mean (Standard Error); unit: percent change
Groups:
- Baseline vs 45-Day Visit: Percentage Changes in Pain Intensity on the Ocular Pain Assessment Survey Between Baseline and the 45-Day Visit after daily ITN
  ITN: Intranasal neurostimulation with TrueTear™ intranasal neurostimulator
- Baseline vs 90-Day Visit: Percentage Changes in Pain Intensity on the Ocular Pain Assessment Survey Between Baseline and the 90-Day Visit after daily ITN
  ITN: Intranasal neurostimulation with TrueTear™ intranasal neurostimulator
Arm/Group | Baseline vs 45-Day Visit | Baseline vs 90-Day Visit
Number analyzed (Participants) | 12 | 6
percent change
  Most eye pain in 24 hours | -31.76 (18.76) | -54.25 (20.55)
  Least eye pain in 24 hours | -12.14 (22.67) | -37.69 (25.46)
  Average eye pain in 24 hours | -30.43 (20.17) | -46.08 (21.35)
  Most eye pain in 2 weeks | -22.89 (18.43) | -43.73 (16.57)
  Least eye pain in 2 weeks | -19.75 (25.93) | -37.50 (26.93)
  Average eye pain in 2 weeks | -24.77 (22.18) | -46.90 (20.85)

9. Secondary Outcome: Overall Percent Change on Impact of Dry Eye in Everyday Life (IDEEL)
Description: IDEEL Quality of Life Questionnaire is a 27-item questionnaire, designed specifically for DED and is divided into three parts. It assesses the quality of life in three aspects of life for the previous 2 weeks: daily activities, work and feelings. The quality of life is assessed on a scale of 0-5, with zero being inability to do the activity. The score is calculated between 0 - 100 with higher scores indicating a better quality of life. Percentage change in IDEEL questionnaire subheading between baseline and day 45 and baseline and day 90 were given below.
Time Frame: Baseline vs day 45 visit and Baseline vs day 90 visit
Population: All patients participated INSTANT visits.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Baseline vs 45 Day Visit: Overall Percent Change on IDEEL questionnaire between baseline and 45 day visit
  IDEEL: Impact of Dry Eye in Everyday Life
  TrueTear™ intranasal neurostimulator (ITN)
  TrueTear™ intranasal neurostimulator (ITN): TrueTear™ intranasal neurostimulator (ITN)
- Baseline vs 90 Day Visit: Overall Percent Change on IDEEL questionnaire between baseline and 90 day visit
  IDEEL: Impact of Dry Eye in Everyday Life
  TrueTear™ intranasal neurostimulator (ITN)
  TrueTear™ intranasal neurostimulator (ITN): TrueTear™ intranasal neurostimulator (ITN)
Arm/Group | Baseline vs 45 Day Visit | Baseline vs 90 Day Visit
Number analyzed (Participants) | 12 | 6
percent change
  Daily Activities | 16.14 (23.72) | 21.83 (17.93)
  Feelings | 17.06 (17.38) | 40.73 (38.43)
  Work | 46.91 (17.82) | 48.80 (40.45)

10. Secondary Outcome: Change in the Intraocular Pressure (IOP) Measured in Each Visit.
Description: Intraocular pressure will be measured by an applanation tonometer used on slit lamp (Goldmann) in mmHg. Change in IOP values between baseline and 90-day is provided below. A healthy eye pressure is between 10 and 21 millimeters of mercury. The differences in intraocular pressure between the baseline and day 45 visits, as well as between the baseline and day 90 visits, are presented below.
Time Frame: Baseline vs day 45 visit and Baseline vs day 90 visit
Population: Patients participated INSTANT study visits.
Measure: Mean (Standard Error); unit: millimeters of mercury (mmHg)
Groups:
- Baseline vs 45 Day Visit: Difference of IOP (intraocular pressure) between baseline and 45 days visits after daily TrueTear™ intranasal neurostimulator (ITN) use.
- Baseline vs 90 Day Visit: Difference of IOP (intraocular pressure) between baseline and 90 days visits after daily TrueTear™ intranasal neurostimulator use.
Arm/Group | Baseline vs 45 Day Visit | Baseline vs 90 Day Visit
Number analyzed (Participants) | 12 | 6
millimeters of mercury (mmHg) | -0.18 (1.10) | -0.43 (0.92)

11. Secondary Outcome: Number of Participants With Adverse Events (Safety)
Description: For safety analyses during the study, patient-reported adverse events that developed after intranasal neurostimulation were recorded.
Time Frame: 90 days
Population: All patients who underwent intranasal neurostimulation were evaluated for safety measures.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: All Patients Who Participated in This Study Were Evaluated for the Safety of ITN
  ITN: TrueTear™ intranasal neurostimulator
Arm/Group | All Patients
Number analyzed (Participants) | 21
Participants
  Migraine Attacks | 2
  Increased Eye Pain | 1
  Increased Facial Pain | 1
  Sinus Irritation and Pain | 1
  Sinus Infection | 1
  Excessive Tearing | 1
  Pain in the nose | 2

12. Secondary Outcome: Number of Participants With Adverse Events (Tolerability)
Description: Tolerability of Intranasal Neurostimulator (ITN) was evaluated by using Ocular Tolerability and Compliance Questionnaire. It assesses symptoms of discomfort in each eye after ITN use.
Time Frame: 90 days
Population: All patients who underwent intranasal neurostimulation and completed Ocular Tolerability and Compliance Questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: All Patients Who Participated in This Study Were Evaluated for the Tolerability of ITN
  ITN: TrueTear™ intranasal neurostimulator (ITN)
Arm/Group | All Patients
Number analyzed (Participants) | 21
Participants
  Eye Itching | 2
  Burning sensation | 3
  Foreign Body Sensation | 2
  Sneezing | 2
  Forehead Throbbing | 1

13. Secondary Outcome: Reduction on Other Concomitant Pain Therapy
Description: After daily intranasal neurostimulation, the change in the number of systemic pain medication between baseline vs 45-day visit and Baseline vs 90-day visit was evaluated.
Time Frame: Baseline vs 45 Day Visit and baseline vs 90 Day Visit
Population: INSTANT patients participated baseline-45 Day Visit and baseline-90 Day Visit
Measure: Mean (Standard Error); unit: Number of medication (n)
Groups:
- Baseline vs 45 Day Visit: Difference in the Number of Systemic Pain Medications Between Baseline and 45-Day Visits After Daily Use of the TrueTear™ Intranasal Neurostimulator
- Baseline vs 90 Day Visit: Difference in the Number of Systemic Pain Medications Between Baseline and 90-Day Visits After Daily Use of the TrueTear™ Intranasal Neurostimulator
Arm/Group | Baseline vs 45 Day Visit | Baseline vs 90 Day Visit
Number analyzed (Participants) | 12 | 6
Number of medication (n) | 0.14 (0.08) | -0.25 (0.25)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Adverse events were collected from patient diaries completed during daily intranasal neurostimulation, verbal reports provided by patients during clinical visits, and patient-completed Ocular Tolerability Questionnaire forms during clinical visits.
Groups:
- All Patients: All patients participated in this study
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 13/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=21)
Excessive tearing (Eye disorders) | 1
Burning Sensation on Eye (Eye disorders) | 3
Foreign Body Sensation on Eye (Eye disorders) | 2
Increased Eye Pain (Eye disorders) | 1
Eye Itching (Eye disorders) | 2
Forehead throbbing (Nervous system disorders) | 1
Migraine Attacks (Nervous system disorders) | 2
Increased Facial Pain (Nervous system disorders) | 1
Pain in the nose (General disorders) | 2
Sinus irritation and Pain (General disorders) | 1
Sinus infection (General disorders) | 1
Sneezing (General disorders) | 2

LIMITATIONS AND CAVEATS:
Patients were not compliant in returning to clinic for follow-up visits. This may be because these visits were to occur on the same day as their routine clinical follow-up visits and the patients repeatedly skipped or cancelled their visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03674892/Prot_SAP_002.pdf
  • Informed Consent Form (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT03674892/ICF_001.pdf